CLINICAL TRIAL: NCT06965166
Title: Pilot Prospective Study of Contrast-Enhanced Photon-Counting Detector CT (PCD-CT) for the Local Staging of Rectal Cancer
Brief Title: Contrast-Enhanced Photon-Counting Detector CT (PCD-CT) for the Local Staging of Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-001797; NCI-2024-10472 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-001797 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-05-01; First posted 2025-05-11 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo PCD-CT on study.
  Interventions: Procedure: PCD-CT

INTERVENTIONS:
Procedure: PCD-CT — Participants undergo PCD-CT scan on study
  Other Names: contrast-enhanced photon-counting detector CT; contrast-enhanced photon-counting detector computed tomography

SUMMARY:
This study evaluates whether images taken using a photon counting detector CT scanner (PCD-CT) can determine the growth of rectal cancer as well as, or better than, MRI for the management of patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 to 99 years of age
* Patients with proven rectal cancer clinically referred for staging pelvic MRI and contrast-enhanced CT of the abdomen and pelvis (for evaluation of liver and peritoneal disease)
* Endoscopic or imaging report that tumor is 2 cm or larger
* Patients who are able and willing to sign the informed consent
* Negative pregnancy test if subject is of child-bearing age (females of child-bearing potential will be screened for pregnancy using a urine pregnancy test, which will be administered by the unit study coordinator at no cost to the patient)

Exclusion Criteria:

* Minors less than 18 years old
* Known mucinous adenocarcinoma (may not enhance well)
* Patient unable to provide written informed consent
* Pregnancy
* estimated Glomerular Filtration Rate (eGFR) ≤ 60
* History of prior moderate or severe contrast reaction including unresponsiveness, severe respiratory distress, convulsions, arrhythmia, cardiopulmonary distress, progressive angioedema, laryngeal edema, dyspnea, bronchospasm, symptomatic tachycardia, symptomatic bradycardia, hypotension, hypertensive crisis
* Any history of premedication prior to iodinated contrast
* Hip replacement/prosthesis
* Patients that consent to participation but do not undergo their clinically indicated MRI scanning for any reason (e.g., bad IV, infiltration, reaction, change in indication)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven rectal cancer clinically referred for staging pelvic MR and contrast-enhanced CT of the abdomen and pelvis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of contrast-enhanced pelvic PCD-CT for CRM involvement | Baseline (after research CT scan has been performed)
  Images from contrast-enhanced pelvic PCD-CT for circumferential resection margin (CRM) involvement will be compared to rectal cancer MRI images. A single-group design will be used to test whether the proportion is non-inferior, with a noninferiority difference (P0 - PB) of -0.1 (H0: P ≤ P0 versus H1: P > P0). The comparison will be made using a one-sided, one-sample exact binomial test, with a Type I error rate (alpha) of 0.05. The limit of non-inferiority will be set at -0.10, meaning that the lower limit of the estimate of the difference between the modalities will be greater than -0.10 for PCD-CT to be non-inferior.

CONTACTS AND LOCATIONS:
Overall Officials: Joel G. Fletcher, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials